CLINICAL TRIAL: NCT05508412
Title: CancerPEP Phase 2 Randomized Trial: Feasibility of a Comprehensive Cancer Patient Empowerment Program Providing Immediate Versus Delayed Stress Reduction Biofeedback Equipment
Brief Title: Cancer Patient Empowerment Program: Phase 2 Feasibility Study
Acronym: CancerPEP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Dalhousie University (Other)
Responsible Party: Principal Investigator, Gabriela Ilie, Associate Professor, Dalhousie University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CancerPEP-Phase2-Protocol
Record Dates: First submitted 2022-08-18; First posted 2022-08-19 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention with HRV monitor (Experimental)
  Interventions: Behavioral: CancerPEP
- Intervention without HRV monitor (Experimental)
  Interventions: Behavioral: CancerPEP

INTERVENTIONS:
Behavioral: CancerPEP — CancerPEP

SUMMARY:
The Cancer Patient Empowerment Program is a comprehensive health promotion program aiming to improve the quality of life as well as both physical and mental health in cancer patients and survivors. The program includes daily email communications over 6 months that encourage strength and aerobic exercise, yoga, stress reduction techniques, dietary improvements, and more.

ELIGIBILITY:
Inclusion Criteria:

* Age >18.
* History of a cancer diagnosis as per the participant's report.
* Safe to exercise and do strength training. Participants who have recovered from a minor stroke or heart condition in the past will require approval from their Family Physician or Cardiologist to participate in the study.
* Participants with advanced cancer (including cancer spread to bones) will need approval from the Study Physician or their Oncologist to participate.
* Existing (or willingness to create) email account and willingness to access email daily.
* Ability to follow website links to watch YouTube videos.
* Ability to understand and speak English.
* Ability to participate in low to moderate levels of physical activity and strength training.
* Ability and willingness to fill out an online survey at baseline, and 6, 12 and possibly 24 months, and a weekly compliance survey for the six months of the program.
* Deemed to have an expected survival greater than 1 year and expected to be well enough to complete the six-month training

Exclusion Criteria:

* Patients deemed unfit to participate in low to moderate level exercise e.g., including but not limited to a myocardial infarction or stroke within the last year, without approval from their Family Physician or Cardiologist that they are safe to exercise.
* Unable to access the internet and lack of a computer or smartphone to receive emails required for study intervention, or unable to click on a link to successfully watch a YouTube video.
* Those with a predicted survival less than 1 year, or not expected to be able to participate in the program for six months.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2022-12-06 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Feasibility (accrual, attrition, compliance, and adverse events) | 6 - 24 months
  As measured by accrual, attrition, compliance rates, and safety by number of adverse events.

SECONDARY OUTCOMES:
Mental Health as assessed by the Kessler Kessler Psychological Distress Scale (K10) | 6 - 24 months
  A 10 item questionnaire that assesses psychological distress. The scale has a score range of 10-50, with higher scores indicating worse mental health.
General Health (Physical and Mental) Quality of Life assessed by the 12-item Short Form Health Survey (SF-12) | 6 - 24 months
  A 12 item questionnaire. The scale has a score range of 0-100, with higher scores indicating better physical and mental health functioning.
Health-Related Quality of Life as assessed by the Functional Assessment of Cancer Therapy - General (FACT-G) | 6 - 24 months
  A 27 item questionnaire that measures the four domains of HRQOL in cancer patients: Physical, social, emotional, and functional well-being. The scale has a score range of 0-108, with higher scores indicating better quality of life.
Personality as assessed by the Ten-Item Personality Inventory (TIPI) | 6 - 24 months
  A 10 item questionnaire assessing the Big-Five personality dimensions (Extraversion, Agreeableness, Conscientiousness, Emotional Stability, Openness to Experiences). The scale has a score range of 1-14 for each dimension with higher scores indicating a higher level of that personality trait.
Alcohol Habit assessed by questions from the NIH Alcohol Consumption questionnaire. | 6 - 24 months
  Questions assessing alcohol consumption
Smoking habit assessed by the Global Adult Tobacco Survey 2020 (GATS). | 6 - 24 months
  Questions assessing smoking use
Diet assessed by the Rapid Eating Assessment for Participants (REAP-S). | 6 - 24 months
  A 16 item questionnaire assessing diet quality. The scale has a score range of 13-39 with a higher score indicating a higher diet quality.
Comorbidity level assessed by the modified Charlson Comorbidity Index (CCI) | 6 - 24 months
  Each category is scored from 1-6. The higher the score, the more likely the predicted outcome will result in mortality or higher resource use.
Availability of social support assessed by the MOS Social Support Survey | 6 - 24 months
  A 19 item questionnaire that assesses emotional/informational support, positive social interaction, tangible support and affectionate support. Higher item scores reflect a higher level of social support.
Sleep Quality as assessed by the Pittsburgh Sleep Quality Index (PSQI) | 6 - 24 months
  A 19 item questionnaire that assesses sleep quality and disturbances. The scale has a score range of 0-21 with a higher score indicating worse sleep quality.
Sedentary behaviour measured by the Sedentary Behaviour Questionnaire (SBQ) for Adults. | 6 - 24 months
  Two 9 item questionnaires (weekday and weekend) with each item scored to none to 6 hours or more. The total score is the sum of the amount of time and as it increases it indicates higher amount of sedentary behaviour.
Sexual functioning in women assessed by the 6-item Female Sexual Function Index (FSFI-6). | 6 - 24 months
  A 6-item shortened version of the original index. Items are rated on a 5-point Likert scale, ranging from 1 to 5, and the other items are rated on a 6-point Likert scale, ranging from 0 to 5. Total scores range from 2 to 30, with lower scores indicating worse sexual functioning.
Sexual functioning in men assessed by the Sexual Health Inventory in Men (SHIM). | 6 - 24 months
  A 5-item questionnaire with scores ranging from 1-25 and lower scores indicating worse sexual functioning.
Anxiety severity assessed by the GAD-7. | 6 - 24 months
  A 7 item questionnaire with scores ranging from 0-21 higher scores indicating more severe level of anxiety.
Relationship satisfaction as assessed by the Dyadic Adjustment Scale (DAS-32). | 6 - 24 months
  A 32 item questionnaire that measure an individual's perceptions of their relationship with an intimate partner. The scale has a total score range of 1-151 with a higher score indicating better satisfaction.
Center for Epidemiologic Studies Depression Scale (CES-D). | 6 - 24 months
  A 20 item questionnaire with a possible range of scores from zero to 60, with the higher scores indicating the presence of more depressive symptomatology.
Satisfaction with Life Scale (SWLS). | 6 - 24 months
  A 5 item questionnaire that was designed to measure subjective well-being. Scores range from 5-35 with higher scores indicating higher satisfaction with life.
Brief Illness Perception Questionnaire (IPQ). | 6 - 24 months
  A 9 item sale that measures an individual's beliefs, feelings, and cognitive representations of one's illness.

CONTACTS AND LOCATIONS:
Locations (1):
- QEII Health Sciences Centre, Halifax, Nova Scotia, Canada

REFERENCES:
- [Derived] Ilie G, Knapp G, Davidson A, Snow S, Dahn HM, MacDonald C, Tsirigotis M, Rutledge RDH. The Cancer Patient Empowerment Program: A Comprehensive Approach to Reducing Psychological Distress in Cancer Survivors, with Insights from a Mixed-Model Analysis, Including Implications for Breast Cancer Patients. Cancers (Basel). 2024 Oct 2;16(19):3373. doi: 10.3390/cancers16193373. PMID 39409993